CLINICAL TRIAL: NCT02737319
Title: A Randomized Trial of Rosuvastatin in Elective Percutaneous Coronary Intervention to Prevent Contrast-induced (CLEAR-CIN).
Brief Title: A Randomized Trial of Rosuvastatin in Elective Angioplasty to Prevent Contrast-induced Nephropathy (CLEAR-CIN).
Acronym: CLEAR-CIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Kleber Bomfim Araujo Martins, MD,PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDPC3851
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Nephropathy
Keywords: Contrast,nephropathy, angioplasty, stable coronary
MeSH Terms: conditions — Kidney Diseases | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Experimental): 40 mg of Rosuvastatin up to 6 hours before elective percutaneous coronary intervention.
  Interventions: Drug: Rosuvastatin
- Control (No Intervention): Use of standard therapy in elective angioplasty.

INTERVENTIONS:
Drug: Rosuvastatin — 40 mg of rosuvastatin before angioplasty
  Other Names: Group 1
  Arms: Rosuvastatin

SUMMARY:
The investigators analyzed the HMG-CoA reductase inhibitor, rosuvastatin, for the prevention of contrast-medium-induced nephropathy in patients undergoing primary angioplasty.

DETAILED DESCRIPTION:
Patients with stable coronary artery disease already taking chronic statin undergoing elective angioplasty are at risk for contrast-medium-induced nephropathy because there are specified risk factors as age more than 75 years, chronic renal insufficiency, diabetes, use of contrast and the lack of effective prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* chronic statin use
* positive stress test findings (electrocardiography, nuclear imaging, or stress echocardiography
* elective angioplasty.

Exclusion Criteria:

* non-statin therapy
* any presentation of ACS within 24 hours before the time of randomization
* current use of potent CYP3A4 inhibitors, including azole antifungals, protease inhibitors, macrolide antibiotics, and cyclosporine
* renal replacement therapy, a history of kidney transplant, pregnant and with renal failure (serum creatinine > 3.0 mg/dl).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Contrast induce nephropathy defined by serum creatinine increase more than 0.3mg/dl or 50% higher than baseline | 48 hours
  Serum creatinine increase more than 0.3mg/dl or 50% higher than baseline

SECONDARY OUTCOMES:
Composite end-point ( all cause of death; acute renal failure and no-fatal mayocardial infarctio. | 48 hours
  Death, myocardial infarction or kidney insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Kleber Bomfim A Martins, MD, PhD, Principal Investigator — Instituto Date Pazzanese de Cardiologia
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No